CLINICAL TRIAL: NCT05464654
Title: VABIP Study (Vaginal Biorevitalization With Polydeoxyribonucleotides) for the Improvement of the Genitourinary Syndrome of Menopause
Brief Title: Vaginal Biorevitalization With Polydeoxyribonucleotides for the Improvement of the Genitourinary Syndrome of Menopause
Acronym: VABIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional 1o de Octubre (Other)
Collaborators: Hospital General Regional No. 1 IMSS (Other Government); Universidad Nacional Autonoma de Mexico (Other); National Polytechnic Institute, Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 012-20170421
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Genitourinary Syndrome of Menopause; Postmenopausal Disorder; Menopause; Vagina Atrophy
Keywords: Polynucleotides; Genitourinary syndrome of menopause; Postmenopause; Vagina atrophy; Vaginal biorevitalization
MeSH Terms: interventions — Drugs, Generic

STUDY DESIGN:
Intervention Model Description: A randomised clinical trial was conducted in 136 postmenopausal women with GSM from the "peri-postmenopause and bone metabolism clinic" of the "Regional Hospital October 1st " of ISSSTE, Mexico, from June to December 2021. The control group (n=64) received local estrogen-based hormonal therapy, applied to the vagina mucosa on Monday, Wednesday, and Friday of each week, for 3 months, while the experimental group (n=72) received local salmon PDRNs on vaginal suppositories, applied solely for six days every night in the first week. The follow-up assessment was done after 3 months.
Who Masked: Outcomes Assessor
Masking Description: The pathologist and colposcopists were blinded to the treatment the participants received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polynucleotide vaginal suppositories (Experimental): In this arm 72 first-time participants of the "peri-postmenopause and bone metabolism clinic" of the "Regional Hospital October 1st " of ISSSTE Mexico, were randomly enrolled to be treated with local salmon polydeoxyribonucleotide (PDRN) therapy.
  Interventions: Drug: 3 g Polynucleotide vaginal suppositories
- Conjugated estrogens cream (Active Comparator): In this arm 64 first-time participants of the "peri-postmenopause and bone metabolism clinic" of the "Regional Hospital October 1st " of ISSSTE Mexico, were randomly enrolled to be treated with the gold-standard treatment with local estrogen-based hormone therapy.
  Interventions: Drug: Conjugated estrogens cream 1g Tube

INTERVENTIONS:
Drug: 3 g Polynucleotide vaginal suppositories — 3 g polynucleotide vaginal suppositories were administered nightly for 6 days.
  Other Names: Tunover®
  Arms: Polynucleotide vaginal suppositories
Drug: Conjugated estrogens cream 1g Tube — Conjugated estrogen cream 1g was applied intravaginally on Monday, Wednesday and Friday for three months.
  Other Names: Generic
  Arms: Conjugated estrogens cream

SUMMARY:
The aim of the study was to compare the efficacy of vaginal biorevitalization to improve the genitourinary syndrome of menopause (GSM) between the gold-standard treatment with local estrogen-based hormone therapy versus local salmon polydeoxyribonucleotide (PDRN) therapy.

DETAILED DESCRIPTION:
The aim of the study was to compare the efficacy of vaginal biorevitalization to improve the genitourinary syndrome of menopause (GSM) between the gold-standard treatment with local estrogen-based hormone therapy versus local salmon polydeoxyribonucleotide (PDRN) therapy. Thus, a randomized clinical trial was conducted in 136 first-time postmenopausal women with GSM, from the "peri-postmenopause and bone metabolism clinic" of the "Regional Hospital October 1st " of the "Institute of Security and Social Services for State Workers (ISSSTE)", from June 2021 to December 2021. Participants were referred by the family medicine service or by another service of the hospital. The control group (n=63) received local estrogen-based hormonal therapy, applied topically to the vagina mucosa on Monday, Wednesday, and Friday of each week, for 3 months, while the experimental group (n=70) received local salmon PDRNs on vaginal suppositories, applied solely for six days every night in the first week. Then, experimental group participants were maintained without further treatment up to the control evaluation. The follow-up assessment was done after 3 months. The alterations in the urogenital domain of the MRS score (items 9-11), vaginal maturity index (VMI), vaginal pH, estrogenic effect, floor pelvic contraction capacity, as well as colposcopy findings, were the main outcomes of the study.

ELIGIBILITY:
Inclusion Criteria:

* First-time patients with the diagnosis of Genitourinary Syndrome of Menopause with an MRS > 5 in the urogenital domain, with alterations in the vaginal maturity index (VMI).

Exclusion Criteria:

* Incomplete clinical records.
* History of prolonged use of steroids.
* Use of alternative local therapies applied in the vagina's mucosa.
* Use of local therapies with vaginal suppositories for any reason 15 days before the beginning of the study.
* Clinical evidence of infectious cervical-vaginitis or vulvovaginitis.
* Evidence of urinary tract infection (UTI).
* Lack of adherence to medical treatment.
* Diagnosis of cancer.
* Diagnosis of depression.
* Diagnosis of uncontrolled primary or secondary immunodeficiencies.
* Allergies to any of the medications administered.
* BIRADS >2 or high risk of developing breast cancer, ovarian cancer or endometrial cancer.
* Use of oral hormonal or non-hormanl therapy.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline urogenital domain score in the Menopause Rating Scale (MRS) at 3 months | 3 months
  Menopause Rating Scale measures the severity of ageing symptoms and their impact on Health-Related Quality of Life. Items 9, 10 and 11 evaluate the urogenital domain. 0 points were considered asymptomatic, 1point indicated mild symptoms, 2-3 points moderate symptoms and > 4 indicated severe symptoms.
Change from baseline Item 9 Menopause Rating Scale (MRS) total score at 3 months | 3 months
  Menopause Rating Scale measures the severity of ageing symptoms and their impact on Health-Related Quality of Life. Item 9 assesses the severity of sexual problems, including changes in libido, sexual activity, and dyspareunia. 0 points were assigned if the participants reported no symptoms, 1 point if they reported mild symptoms, 2 points if they reported moderate symptoms, 3 points if they reported severe symptoms, and 4 points if they reported extremely severe symptoms.
Change from baseline Item 10 Menopause Rating Scale (MRS) total score at 3 months | 3 months
  Menopause Rating Scale measures the severity of ageing symptoms and their impact on Health-Related Quality of Life. Item 10 assesses the severity of urinary problems such as polyuria, urinary urgency, bladder instability, and urinary incontinence. 0 points were assigned if the participants reported no symptoms, 1 point if they reported mild symptoms, 2 points if they reported moderate symptoms, 3 points if they reported severe symptoms, and 4 points if they reported extremely severe symptoms.
Change from baseline Item 11 Menopause Rating Scale (MRS) total score at 3 months | 3 months
  Menopause Rating Scale measures the severity of ageing symptoms and their impact on Health-Related Quality of Life. Item 11 assesses the severity of vaginal dryness. 0 points were assigned if the participants reported no symptoms, 1 point if they reported mild symptoms, 2 points if they reported moderate symptoms, 3 points if they reported severe symptoms, and 4 points if they reported extremely severe symptoms.
Change from baseline Vaginal Maturity Index (VMI) at 3 months | 3 months
  The vaginal maturation index (VMI) is used to assess the hormonal status of the vaginal epithelium, which quantifies the proportions of cell types in the vaginal epithelium. The VMI was evaluated through vaginal cytology, where the percentage of basal/parabasal, intermediate and superficial cells were calculated.
Change from baseline Estrogenic Effect at 3 months | 3 months
  The estrogenic effect is used to evaluate the local action of estrogens in the vaginal epithelium. The higher value, it means that it is having a greater trophic effect due to local estrogen stimulation. To calculate this outcome, it was used the next formula:
  Estrogenic effect= [(% of basal/parabasal cells*0)+(% of intermediate cells*0.5)+(% of superficial cells*1)]
Change from baseline Oxford grading scale at 3 months | 3 months
  The Oxford grading scale evaluates the contraction capacity of the muscles of the pelvic floor. It was used at the time of vaginal examination. 0 points meant no contraction , 1 point a flicker contraction, 2 points a weak contraction, 3 points a moderate contraction, 4 points a good contraction, and 5 points a strong contraction.
Change from baseline vaginal pH at 3 months | 3 months
  Vaginal pH tests measure the acidity of the vagina. A normal vaginal pH value was considered when it was between 4.0 and 5.
Change from baseline colposcopic findings at 3 months | 3 months
  The presence or absence of vaginal folds, paleness and vaginal lesions were colposcopic findings that were evaluated as nominal dichotomous variables. Lugol's staining was performed during colposcopy. The degree of Lugol's staining was evaluated as an ordinal variable with 4 degrees, depending on the intensity of staining of the vaginal mucosa.

CONTACTS AND LOCATIONS:
Overall Officials: Juan M Ocampo-Godinez, M.D., Ph.D., Study Director — Laboratorio de Bioingenieria de Tejidos, UNAM; Patricia Loranca-Moreno, M.D., M.Sc., Principal Investigator — Hospital Regional 1o de Octubre, ISSSTE
Locations (1):
- Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE, Mexico City, Mexico

REFERENCES:
- [Background] The NAMS 2020 GSM Position Statement Editorial Panel. The 2020 genitourinary syndrome of menopause position statement of The North American Menopause Society. Menopause. 2020 Sep;27(9):976-992. doi: 10.1097/GME.0000000000001609. PMID 32852449
- [Background] Schneider HP, Heinemann LA, Rosemeier HP, Potthoff P, Behre HM. The Menopause Rating Scale (MRS): reliability of scores of menopausal complaints. Climacteric. 2000 Mar;3(1):59-64. doi: 10.3109/13697130009167600. PMID 11910611
- [Background] Heinemann K, Assmann A, Mohner S, Schneider HP, Heinemann LA. [Reliability of the Menopause Rating Scale (MRS): Investigation in the German population]. Zentralbl Gynakol. 2002 Mar;124(3):161-3. doi: 10.1055/s-2002-32268. German. PMID 12070795
- [Background] Schneider HP, Rosemeier HP, Schnitker J, Gerbsch S, Turck R. Application and factor analysis of the menopause rating scale [MRS] in a post-marketing surveillance study of Climen. Maturitas. 2000 Dec 29;37(2):113-24. doi: 10.1016/s0378-5122(00)00177-8. PMID 11137330
- [Background] Heinemann K, Ruebig A, Potthoff P, Schneider HP, Strelow F, Heinemann LA, Do MT. The Menopause Rating Scale (MRS) scale: a methodological review. Health Qual Life Outcomes. 2004 Sep 2;2:45. doi: 10.1186/1477-7525-2-45. PMID 15345062
- [Background] Weber MA, Limpens J, Roovers JP. Assessment of vaginal atrophy: a review. Int Urogynecol J. 2015 Jan;26(1):15-28. doi: 10.1007/s00192-014-2464-0. Epub 2014 Jul 22. PMID 25047897
- [Background] McCracken JM, Balaji S, Keswani SG, Hakim JC. An Avant-Garde Model of Injury-Induced Regenerative Vaginal Wound Healing. Adv Wound Care (New Rochelle). 2021 Apr;10(4):165-173. doi: 10.1089/wound.2020.1198. Epub 2020 Aug 10. PMID 32602816
- [Background] Chung HS, Lee HS, Park K. Estrogen modulates epithelial progenitor cells in rat vagina. Investig Clin Urol. 2021 May;62(3):349-353. doi: 10.4111/icu.20200513. Epub 2021 Apr 2. PMID 33834644
- [Background] Rahn DD, Carberry C, Sanses TV, Mamik MM, Ward RM, Meriwether KV, Olivera CK, Abed H, Balk EM, Murphy M; Society of Gynecologic Surgeons Systematic Review Group. Vaginal estrogen for genitourinary syndrome of menopause: a systematic review. Obstet Gynecol. 2014 Dec;124(6):1147-1156. doi: 10.1097/AOG.0000000000000526. PMID 25415166
- [Background] Nappi RE, Martini E, Cucinella L, Martella S, Tiranini L, Inzoli A, Brambilla E, Bosoni D, Cassani C, Gardella B. Addressing Vulvovaginal Atrophy (VVA)/Genitourinary Syndrome of Menopause (GSM) for Healthy Aging in Women. Front Endocrinol (Lausanne). 2019 Aug 21;10:561. doi: 10.3389/fendo.2019.00561. eCollection 2019. PMID 31496993
- [Result] The NAMS 2017 Hormone Therapy Position Statement Advisory Panel. The 2017 hormone therapy position statement of The North American Menopause Society. Menopause. 2017 Jul;24(7):728-753. doi: 10.1097/GME.0000000000000921. PMID 28650869